CLINICAL TRIAL: NCT02922140
Title: The Impact of Pharmaceutical Care Practice on Patients in Cardiac Rehabilitation Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, eman ahmed el-said casper, Teaching Assisstant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHCL49
Record Dates: First submitted 2016-09-20; First posted 2016-10-04 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Acute Coronary Syndrome
Keywords: pharmaceutical care service, clinical pharmacist; Cardiac rehabilitation unit; Acute coronary syndrome; patient education and counselling
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): will receive standard care by physician in attendance
- intervention group (Active Comparator): will be supplied by clinical pharmaceutical care services provided by the clinical pharmacist plus standard care by physician in attendance.
  Interventions: Behavioral: pharmaceutical care service

INTERVENTIONS:
Behavioral: pharmaceutical care service
  Other Names: pharmaceutical care plan; Comprehensive health care services
  Arms: intervention group

SUMMARY:
This study aims to investigate the role of clinical pharmacist in the development of a pharmaceutical care program for patients with Acute coronary syndrome tailored to their specific learning needs and their cultural context, and to verify the program's effects on physiological factors and recurrent symptoms or cardiac events.

ELIGIBILITY:
Inclusion Criteria:

1. Are diagnosed with Acute coronary syndrome (ischemic heart disease) by their primary cardiologist, treated with medication, percutaneous coronary angioplasty, or coronary artery bypass graft.
2. At 20-79 years of age.
3. Has the ability to perform regular physical activity according to the patients' self-identification and the judgment of their primary cardiologist.
4. Willing to participate in this study.
5. Able to be reached by telephone postdischarge.

Exclusion Criteria:

1. Patients with cognitive impairment.
2. If they need professional help to take their medication at home.
3. With terminal illness.
4. Inability to communicate.
5. Severe arrhythmia.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in the level of patient education about disease, drugs and lifestyle modification using coronary artery disease education questionnaire (CADE-Q) | three months
  at baseline and after three months
Change in the number of solved drug-related problems | three months
  assessment of drug-related problems at baseline and solving them during three months
Assessment of medications adherence: (Eight-item Morisky adherence questionnaire). | three months
  at baseline and after three months

SECONDARY OUTCOMES:
Assessment of quality of life: (36-items self-care Health survey (SF-36)). | three months
  at baseline and after three months
Assessment of smoker's dependence on cigarette smoking: (using the Fagerstrom Test for Nicotine Dependence). | three months
  at baseline and after three months
Change in heart rate [HR] (Bpm). | three months
  at baseline and after three months
Change in Lipid profile : total cholesterol (mg/dl), triglycerides(mg/dl), and low density lipoprotein cholesterol(mg/dl), high density lipoprotein (mg/dl) | three months
  at baseline and after three months
Change in levels of fasting blood glucose (mg/dl) | three months
  at baseline and after three months
Change in systolic and diastolic blood pressure [BP] (mmHg). | three months
  at baseline and after three months

OTHER OUTCOMES:
Change in potassium (mmol/l). | three months
  at baseline and after three months
Change in sodium (mmol/l). | three months
  at baseline and after three months
Change in serum creatinine (mg/dl). | three months
  at baseline and after three months
Change in waist circumference (cm). | three months
  at baseline and after three months
Change in Liver function tests: aspartate aminotransferase enzyme (AST) (u/l), alanine aminotransferase (ALT) (u/l) | three months
  at baseline and after three months
Change in Kidney function tests : serum urea (mg/dl). | three months
  at baseline and after three months
Change in anthropometric measurements (body mass index [BMI] (Kg/m^2)) | three months
  at baseline and after three months

CONTACTS AND LOCATIONS:
Overall Officials: Eman A. Casper, bachelor, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmed Casper E, Mohmed El Wakeel L, Ayman Saleh M, Hamed El-Hamamsy M. The impact of a comprehensive pharmaceutical care intervention in addition to cardiac rehabilitation program on outcomes of post-acute coronary syndrome patients: A pilot study. Patient Educ Couns. 2022 Oct;105(10):3164-3168. doi: 10.1016/j.pec.2022.06.004. Epub 2022 Jun 10. PMID 35701314